CLINICAL TRIAL: NCT00327990
Title: A Multi Centre, Randomised, Open Label, Cross-over Study to Evaluate the Percentage of False Negative Osteoporosis Diagnosis's Using the Standard Case-finding Procedure as Described by the Dutch Institute for Healthcare (CBO) and to Determine the Preference of Adult Osteoporosis Patients Between Once Monthly Dosing of Ibandronate (150 mg) and Once Weekly Dosing of Alendronate (70 mg)
Brief Title: Evaluation Of Missed Osteoporosis Diagnoses, And Preference Between Once Monthly Ibandronate And Once Weekly Alendronate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IBN104125
Record Dates: First submitted 2006-05-18; First posted 2006-05-19 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Osteoporosis
Keywords: ibandronate; osteoporosis; preference; case-finding; post-menopausal; alendronate
MeSH Terms: conditions — Osteoporosis | interventions — Ibandronic Acid; Alendronate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ibandronate
Drug: Alendronate
  Other Names: Ibandronate

SUMMARY:
This is a two part study (screening and treatment). The first part (screening) is designed to evaluate the percentage of patients missed in diagnosing osteoporosis by general practitioners (GP's). The second part (treatment) is designed to determine the preference by patients for the once monthly ibandronate or the once weekly alendronate.

DETAILED DESCRIPTION:
A multi-centre, randomised, open-label, cross-over study to evaluate the percentage of false negative osteoporosis diagnoses using the standard case-finding procedure as described by the Dutch Institute for Health Care (CBO) and to determine the preference of adult osteoporosis patients between once monthly dosing of ibandronate (150 mg) and once weekly dosing of alendronate (70 mg).

ELIGIBILITY:
Inclusion Criteria:

* Women registered with a GP, without a prior history of osteoporosis. According to a case-finding procedure, osteoporosis will be diagnosed or excluded.

Exclusion criteria:

* Abnormalities of the esophagus which delay esophageal emptying such as stricture or achalasia.
* Inability to stand or sit in the upright position for 60 minutes.
* Previous use of bone active agents (e.g. strontium, PTH).
* Significant medical condition which may preclude the patient's ability to complete the study.
* History of alcohol or drug abuse.
* Hypersensitivity to any component of the bisphosphonates alendronate and ibandronate.
* Administration of any investigational drug within 30 days preceding the first dose of the study drug.
* Serum total calcium > 10.5 mg/dL or < 8.0 mg/dL (equivalent to 2.63 mmol/L and 1.99 mmol/L).
* Osteoporosis by secondary causes, will be excluded especially when an isolated deformity of the vertebral body is detected during x-ray analysis.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2005-04; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Part 1: Percentage of patients falsely not diagnosed with osteoporosis using the standard case-finding and additional X-ray procedure in GP practice. Part 2: Patient preference for once monthly ibandronate or once weekly alendronate

SECONDARY OUTCOMES:
Part 1: To assess the safety and tolerance of both ibandronate and alendronate. Part 2: To assess patient preference in reminder methods during once monthly ibandronate regimen: postcard, text message or telephone patient relationship program.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (36):
- Netherlands (36):
  - GSK Investigational Site, Bennebroek
  - GSK Investigational Site, Breda
  - GSK Investigational Site, Damwoude
  - GSK Investigational Site, Driebergen-Rijsenburg
  - GSK Investigational Site, Eersel
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Enschede
  - GSK Investigational Site, Etten-Leur
  - GSK Investigational Site, Geleen
  - GSK Investigational Site, Groesbeek
  - GSK Investigational Site, Heerlen
  - GSK Investigational Site, Hengelo
  - GSK Investigational Site, Hoogvliet
  - GSK Investigational Site, Hoogwoud
  - GSK Investigational Site, Hulst
  - GSK Investigational Site, Landgraaf
  - GSK Investigational Site, Losser
  - GSK Investigational Site, Midwoud
  - GSK Investigational Site, Nijverdal
  - GSK Investigational Site, Nunspeet
  - GSK Investigational Site, Oldebroek
  - GSK Investigational Site, Oosterend
  - GSK Investigational Site, Oudenbosch
  - GSK Investigational Site, Poortvliet
  - GSK Investigational Site, Prinsenbeek
  - GSK Investigational Site, Raalte
  - GSK Investigational Site, Ridderkerk
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Spijkenisse
  - GSK Investigational Site, The Hague
  - GSK Investigational Site, Tilburg
  - GSK Investigational Site, Voerendaal
  - GSK Investigational Site, Wassenaar
  - GSK Investigational Site, Wildervank
  - GSK Investigational Site, Woerden
  - GSK Investigational Site, Zaandam